CLINICAL TRIAL: NCT04261673
Title: A Randomised Controlled Trial to Evaluate Decompressive Craniectomy for Patients With Cerebral Herniation Undergoing Evacuation of Acute Epidural Hematoma
Brief Title: Prospective Randomized Evaluation of Decompressive Ipsilateral Craniectomy for Traumatic Acute Epidural Hematoma
Acronym: PREDICT-AEDH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Shenzhen Second People's Hospital (Other); Clinical Research Institute, Shanghai Jiao Tong University School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREDICT-AEDH
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Epidural Hematoma; Brain Herniation; Decompressive Craniectomy; Craniotomy
MeSH Terms: conditions — Hematoma, Epidural, Spinal | interventions — Decompressive Craniectomy; Craniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompressive Craniectomy (Experimental): After the evacuation of epidural hematoma, the bone flap should not be replaced at the end of the operation.
  Interventions: Procedure: Decompressive Craniectomy
- Craniotomy (Experimental): After the evacuation of epidural hematoma, the bone flap must be replaced and fixed with an appropriate fixation system.
  Interventions: Procedure: Craniotomy

INTERVENTIONS:
Procedure: Decompressive Craniectomy — A large bone flap must be raised. The evacuation of epidural hematoma is depended on surgeon's preference. The bone flap should not be replaced at the end of the operation. DC has an advantage in controlling brain swelling, but patient is necessary to have another operation of cranioplasty to reconstruct the skull in the future.
  Arms: Decompressive Craniectomy
Procedure: Craniotomy — A large bone flap must be raised. The evacuation of epidural hematoma is depended on surgeon's preference. However, the bone flap must be replaced and fixed with fixation system (plates and screws). The patient will not need an additional operation to rebuild the skull in the future. But undisciplinable brain swelling and increased intracranial pressure may happen in some patients, and additional decompressive craniectomy is recommended in these cases.
  Arms: Craniotomy

SUMMARY:
Although craniotomy provides a more complete evacuation of the acute epidural hematoma, there are insufficient data to support specific surgical treatment method. We aim to perform a multi-center, parallel-group randomized clinical trial to compare the outcome and cost-effectiveness of decompressive craniectomy versus craniotomy for the treatment of traumatic brain injury patients with cerebral herniation undergoing evacuation of an acute epidural hematoma.

DETAILED DESCRIPTION:
The incidence of epidural hematoma (EDH) among traumatic brain injury (TBI) patients has been reported to be in the range of 2.7 to 4%. Among patients in coma, up to 9% harbored an EDH requiring craniotomy. The mortality in patients in all age groups and GCS scores undergoing surgery for evacuation of EDH is approximately 10%. The decision to operate on an acute EDH (AEDH) is usually based on the patient's GCS score, age, pupillary abnormalities, comorbidities, CT findings, associated intracranial lesions, in delayed decisions, the time between neurological deterioration and surgery, and intracranial pressure. An AEDH greater than 30 ml should be surgically evacuated regardless of the patient's Glasgow Coma Scale (GCS) score. There are insufficient data to support one surgical treatment method. However, craniotomy provides a more complete evacuation of the hematoma for patients with an AEDH that require an operation to remove the clot. But whether decompressive craniectomy (DC) should be employed still has considerable controversy. The choice of operative technique is influenced by the surgeon's expertise, training, and evaluation of a particular situation. The difference between these two procedures is that a bone flap is left out before closing the skin in DC. Both approaches are widely used among neurological surgeons (although the indications may differ), therefore there is sufficient experience in the centers to set up a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Clear medical history of traumatic brain injury;
2. Within 12 hours after injury;
3. Unilateral mydriasis or bilateral mydriasis before the operation;
4. Acute supratentorial epidural hematoma and signs of brain stem compression on CT scan, representing the leading cause of operation, despite any other minor intracranial injuries associated (e.g., subarachnoid hemorrhage and contusion);
5. The admitting neurosurgeon considers that the epidural hematoma needs to be evacuated with a craniotomy or decompressive craniectomy.
6. With informed consent.

Exclusion Criteria:

1. Previous intracranial surgery prior to trauma;
2. Patients with a score of 3 on the GCS, with bilateral fixed and dilated pupils, bleeding diathesis or defective coagulation, or other injuries that were deemed to be unsurvivable;
3. Patients who had injury of the oculomotor nerve;
4. Patients are considered to be operated mainly by following pathological change on CT: subdural hematoma, intracerebral hemorrhage, large size infarction, et al., but not because of epidural hematoma;
5. Severe pre-existing disability or severe co-morbidity which would lead to a poor outcome even if the patient is supposed to a good recovery from the TBI;
6. Pregnant female.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-05-23 (Actual); Primary Completion 2025-09-14 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
GOSE (extended Glasgow Outcome Scale) scores | 6 months post-injury
  The primary outcome is indicated by the long-term functional outcomes, including overall mortality and the score on the "Extended Glasgow Outcome Scale" (GOS-E). "Extended Glasgow Outcome Scale" is the unabbreviated scale title, minimum value is 1 and maximum value is 8, which was scored as follows and higher scores mean a better outcome:
  1. death;
  2. persistent vegetative state;
  3. lower severe disability;
  4. upper severe disability (stratum 3 and 4 were considered as severe disability, with permanent requirement for help with daily living);
  5. lower moderate disability;
  6. upper moderate disability (stratum 5 and 6 were considered as mild disability, without a need for assistance in everyday life, that might, however, require special equipment for employment);
  7. lower good recovery;
  8. upper good recovery (stratum 7 and 8 were considered as good recovery).

SECONDARY OUTCOMES:
incidence of post-operative cerebral infarction | within 6 months post-injury
  Patients have clinical deterioration after an initial surgery because of post-operative cerebral infarction.
incidence of additional craniocerebral surgery | within 6 months post-injury
  Patients have additional craniocerebral surgical operation as a result of clinical deterioration.
length of stay in hospital | within 6 months post-injury
  The length of patient's stay in hospital after initial surgery, which must due to AEDH related medical treatment. Number of days in hospital are used to evaluate length, and patients with poor treatment effect may need longer hospital stays.
detailed economic evaluation | within 6 months post-injury
  Total medical expense related to treatment of AEDH, including the costs of operations, hospitalization and rehabilitation. Different operations have different medical expense，and patients with poor treatment effect may need more medical expense. We record and evaluate the total medical expense of the entire AEDH treatment process, within 6 months post-injury.
incidence of serious adverse events | within 6 months post-injury
  Serious adverse events (SAE) is defined as an untoward occurrence that:
  1. results in death;
  2. is life-threatening;
  3. requires hospitalization or prolongation of existing hospitalization;
  4. results in persistent or significant disability or incapacity;
  5. is otherwise considered medically significant by the investigator.
quality of life (EQ-5D-5L) | at 1,3 and 6 months post-injury
  Unabbreviated scale title is "5-level EuroQol five dimensions" questionnaire. The EQ-5D is a generic instrument for describing and valuing health. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
MMSE (mini-mental state examination) scores | at 1,3 and 6 months post-injury
  Unabbreviated scale title is "mini-mental state examination", and minimum value is 0 and maximum value is 30. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Junfeng Feng, MD, Principal Investigator — Department of Neurosurgery,Renji Hospital,School of Medicine,Shanghai Jiao Tong University
Locations (1):
- Department of Neurosurgery, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bullock MR, Chesnut R, Ghajar J, Gordon D, Hartl R, Newell DW, Servadei F, Walters BC, Wilberger JE; Surgical Management of Traumatic Brain Injury Author Group. Surgical management of acute epidural hematomas. Neurosurgery. 2006 Mar;58(3 Suppl):S7-15; discussion Si-iv. PMID 16710967
- [Background] Li LM, Kolias AG, Guilfoyle MR, Timofeev I, Corteen EA, Pickard JD, Menon DK, Kirkpatrick PJ, Hutchinson PJ. Outcome following evacuation of acute subdural haematomas: a comparison of craniotomy with decompressive craniectomy. Acta Neurochir (Wien). 2012 Sep;154(9):1555-61. doi: 10.1007/s00701-012-1428-8. Epub 2012 Jun 30. PMID 22752713
- [Background] Lin H, Wang WH, Hu LS, Li J, Luo F, Lin JM, Huang W, Zhang MS, Zhang Y, Hu K, Zheng JX. Novel Clinical Scale for Evaluating Pre-Operative Risk of Cerebral Herniation from Traumatic Epidural Hematoma. J Neurotrauma. 2016 Jun 1;33(11):1023-33. doi: 10.1089/neu.2014.3656. Epub 2016 Jan 28. PMID 25393339
- [Background] Wang WH, Hu LS, Lin H, Li J, Luo F, Huang W, Lin JM, Cai GP, Liu CC. Risk factors for post-traumatic massive cerebral infarction secondary to space-occupying epidural hematoma. J Neurotrauma. 2014 Aug 15;31(16):1444-50. doi: 10.1089/neu.2013.3142. Epub 2014 Jun 25. PMID 24773559
- [Derived] Yang C, Huang X, Feng J, Xie L, Hui J, Li W, Jiang J. Prospective Randomized Evaluation of Decompressive Ipsilateral Craniectomy for Traumatic Acute Epidural Hematoma (PREDICT-AEDH): study protocol for a randomized controlled trial. Trials. 2021 Jun 29;22(1):421. doi: 10.1186/s13063-021-05359-6. PMID 34187537